CLINICAL TRIAL: NCT01514227
Title: Nobori Dual Antiplatelet Therapy as Appropriate Duration.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Associations for Establishment of Evidence in Interventions (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIPPON 5.0
Record Dates: First submitted 2011-12-22; First posted 2012-01-23 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Aspirin; thienopyridine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Short-term DAPT (6 months) group (Experimental): 6 months DAPT (aspirin and thienopyridine) prescription following Nobori stent
  Interventions: Drug: Aspirin or thienopyridine
- Long-term DAPT (18 months) group (Experimental): 18 months DAPT (aspirin and thienopyridine) prescription following Nobori stent
  Interventions: Drug: Aspirin and thienopyridine

INTERVENTIONS:
Drug: Aspirin or thienopyridine — Subjects randomized 6 month DAPT will be prescribed either aspirin or thienopyridine (clopidogrel or ticlopidine) following 6 months DAPT for the duration of study, which is left on the physician's discretion.
  Arms: Short-term DAPT (6 months) group
Drug: Aspirin and thienopyridine — Subjects randomized 18 month DAPT will be prescribed both aspirin and thienopyridine (clopidogrel or ticlopidine) for 18 month after stenting.
  Arms: Long-term DAPT (18 months) group

SUMMARY:
NIPPON trial is a prospective, randomized, trial comparing 6 and 18 months Dual Antiplatelet Therapy (DAPT) following Nobori stent deployment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects > 20 years old
* Undergoing percutaneous intervention with Nobori deployment
* No contraindication to prolonged DAPT

Exclusion Criteria:

* Subjects absolutely necessitating continuous DAPT
* Planned surgery necessitating discontinuation of antiplatelet therapy after enrollment.
* Active pathological bleeding
* Status of cardiogenic shock at enrollment
* Pregnant women
* Life expectancy of < 1.5 years
* Subjects unable to give informed consent
* Episode of stroke < 6 months
* Subjects with allergies or hypersensitivity to material of coating, Biolimus A9, and antiplatelet drugs.
* Subjects treated with other kind of DES or BMS during the index procedure
* Previous intervention with DES < 6 months.
* Study participation impractical per investigator judgment

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3773 (Actual)
Dates: Start 2011-12; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Net adverse clinical and cerebral event (NACCE) | 18 months
  NACCE include all-cause death, non-fatal myocardial infarction, cerebrovascular events, and major bleeding.

SECONDARY OUTCOMES:
All-cause death | 18 months
Non-fatal myocardial infarction | 18 months
Cerebrovascular events | 18 months
Major bleeding | 18 months
Rate of target lesion revascularization | 18 months
Minor bleeding | 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Non-profit organization Associations for Establishment of Evidence in Interventions, Minato-ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nakamura M, Iijima R, Ako J, Shinke T, Okada H, Ito Y, Ando K, Anzai H, Tanaka H, Ueda Y, Takiuchi S, Nishida Y, Ohira H, Kawaguchi K, Kadotani M, Niinuma H, Omiya K, Morita T, Zen K, Yasaka Y, Inoue K, Ishiwata S, Ochiai M, Hamasaki T, Yokoi H; NIPPON Investigators. Dual Antiplatelet Therapy for 6 Versus 18 Months After Biodegradable Polymer Drug-Eluting Stent Implantation. JACC Cardiovasc Interv. 2017 Jun 26;10(12):1189-1198. doi: 10.1016/j.jcin.2017.04.019. PMID 28641838